CLINICAL TRIAL: NCT03270670
Title: A Pilot Study Evaluating the Performance of 19-gauge Needles in Testing Molecular Markers in Samples Obtained Via Endobronchial Ultrasound Guided Needle Aspiration of Lymph Nodes in Patients With Lung Cancer
Brief Title: Olympus - 19-gauge Needle
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00082253
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to test whether the 19-gauge needle can collect more tissue and get better sampling during a bronchoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known or suspected lung cancer with mediastinal adenopathy as defined by a mediastinal lymph node >0.5 cm in short axis on EBUS or any lymph node with uptake on FDG-PET scan that is higher than background PET activity.
* Participants must lack bleeding disorders

Exclusion Criteria:

* Subjects who lack fitness for flexible bronchoscopy as determined by the physician performing the bronchoscopy before the procedure
* Subjects with suspected sarcoidosis, lymphoma, or metastatic cancer from other sites (i.e. those without a known or suspected lung primary)
* Subjects on anticoagulation (other than Aspirin) whom cannot have their anticoagulation held for the procedure due to other clinical reasons (i.e. recent cardiac stent placement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing a standard of care bronchoscopy to determine lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Molecular marker test | Day of Procedure
  Descriptive statistics will be used to calculate the success rate of the procedure in successful performance of molecular marker testing

CONTACTS AND LOCATIONS:
Overall Officials: Momen Wahidi, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - Duke Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No